CLINICAL TRIAL: NCT06439212
Title: Assessing the Efficacy of Ginger Powder Capsules as an Analgesic for Intraoperative and Post- Endodontic Pain Management in Mandibular Molars With Symptomatic Irreversible Pulpitis: A Randomized Controlled Trial
Brief Title: the Efficacy of Ginger Powder as an Analgesic for Intraoperative and Post- Endodontic Pain Management
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Alderbashi, Master degree student - Department of Endodontics - Faculty of Dentistry - Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ginger as an Analgesic for EPM
Record Dates: First submitted 2024-05-18; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Endodontic Disease
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ginger (Experimental): Choosing ginger as a pain analgesic is significant due to its anti-inflammatory properties. The presence of active compounds, like shogaols, suggests ginger could provide a clinically effective and safer alternative in managing intra-operative and post-endodontic pain.
  Patient will receive one capsule of 500mg ginger powder capsule thrice daily for two days. First dose will be administered 1 hour before starting endodontic treatment.
  Interventions: Drug: Ginger powder capsule
- Placebo (Placebo Comparator): Patient will receive one capsule of placebo thrice daily for two days. First dose will be administered 1 hour before starting endodontic treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ginger powder capsule — Patient will receive one capsule of 500mg ginger powder capsule thrice daily for two days. First dose will be administered 1 hour before starting endodontic treatment.
  Arms: Ginger
Drug: Placebo — Patient will receive one capsule of placebo thrice daily for two days. First dose will be administered 1 hour before starting endodontic treatment.
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the analgesic effect of ginger powder capsules compared to placebo on intra-operative and post-operative pain of single-visit endodontic treatment of mandibular molars with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
The pharmacological pain management usually includes administration of systemic analgesics, anti-inflammatory drugs, or antibiotics drugs. The inhibition of the inflammatory process is one of the methods to reduce or prevent pain during and after treatment.

Ginger has a lengthy history of use as a herbal medicine. Ginger has been used in traditional Chinese and Indian medicine to treat a variety of diseases, including arthritis, stomachaches, diarrhea, nausea, asthma, and respiratory problems. It was discovered that ginger also contains substances that prevent PG production. This discovery gave its anti-inflammatory benefits a solid scientific justification. Following research, it was discovered that some of the components of ginger share pharmacological traits with a novel family of dual-acting NSAIDs. These substances have significantly fewer adverse effects than traditional NSAIDs and can inhibit arachidonic acid metabolism via both the cyclooxygenase (COX) and lipoxygenase (LOX) pathways.

Various animal studies have shown that taking dried ginger or ginger extract orally can decrease acute inflammation. Numerous clinical studies back up the effectiveness of ginger in treating osteoarthritis, and in some instances, a noticeable decrease in knee pain has been reported. In some of these studies, it was discovered that ginger, even when used for extended amounts of time, significantly reduced pain and swelling in patients with osteoarthritis, rheumatoid arthritis, and muscular pain.

There have been no studies done to evaluate the impact of ginger powder on intra and post-endodontic pain. In order to find the effects of ginger powder capsules on pain after endodontic treatment, the current study was performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aging between 18-45 years old.
2. Patients with mandibular molar with signs and symptoms of symptomatic irreversible pulpitis.
3. Systemically- healthy patients (ASA I or II).
4. Patients who agree to attend for recall appointments.
5. Patients who can understand pain scale and can sign the informed consent.

Exclusion Criteria:

1. Pregnant or lactating female patients.
2. Patients allergic to ginger, articaine or any other medicament material used in the study.
3. History of peptic ulceration.
4. Periapical abscess or fistula.
5. Non-restorable teeth.
6. Moderate or severe marginal periodontitis i.e. pocket probe>3mm.
7. Patients on Aspirin, Clopidogrel, Dalteparin and Warfarin.
8. Radiographic evidence of external or internal root resorption vertical root fracture, perforation, calcification.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | Pain will be assessed at 6 hours, 12 hours, 24 hours and 48 hours postoperatively
  Pain will be assessed using Heft-Parker visual analog scale (HP-VAS). HP-VAS is an 170 mm scale consisting of numbers from 0 to 170. 0 readings represent "no pain"
  1- 54 readings represent "mild pain" 55 - 114 readings represent "moderate pain" 115 - 170 readings represent "severe pain" No to mild pain will be considered as effective medication while moderate to severe pain will be regarded as not effective medication.

SECONDARY OUTCOMES:
Intraoperative pain | Pain will be assessed during the procedure
  Pain will be assessed using Heft-Parker visual analog scale (HP-VAS). HP-VAS is an 170 mm scale consisting of numbers from 0 to 170. 0 readings represent "no pain"
  1- 54 readings represent "mild pain" 55 - 114 readings represent "moderate pain" 115 - 170 readings represent "severe pain" No to mild pain will be considered as effective medication while moderate to severe pain will be regarded as not effective medication.
Rescue-analgesic intake by the patient after endodontic treatment. | Taken after 48 hours post-operatively
  The patient will be asked if they needed a rescue analgesic or not, when and how many times.

REFERENCES:
- [Background] Menon P, Perayil J, Fenol A, Rajan Peter M, Lakshmi P, Suresh R. Effectiveness of ginger on pain following periodontal surgery - A randomized cross-over clinical trial. J Ayurveda Integr Med. 2021 Jan-Mar;12(1):65-69. doi: 10.1016/j.jaim.2020.05.003. Epub 2020 Jul 2. PMID 32624375
- [Background] Rayati F, Hajmanouchehri F, Najafi E. Comparison of anti-inflammatory and analgesic effects of Ginger powder and Ibuprofen in postsurgical pain model: A randomized, double-blind, case-control clinical trial. Dent Res J (Isfahan). 2017 Jan-Feb;14(1):1-7. doi: 10.4103/1735-3327.201135. PMID 28348610
- [Background] Alshibani N, Al-Kattan R, Alssum L, Basudan A, Shaheen M, Alqutub MN, Al Dahash F. Postoperative Analgesic and Anti-inflammatory Effectiveness of Ginger (Zingiber officinale) and NSAIDs as Adjuncts to Nonsurgical Periodontal Therapy for the Management of Periodontitis. Oral Health Prev Dent. 2022 Jul 13;20:227-232. doi: 10.3290/j.ohpd.b3125633. PMID 35695692